CLINICAL TRIAL: NCT03322189
Title: Medical Provider Experience and Assessment on Documenting Prescribing and Plan of Care Changes Due to Pharmacogenomics Testing
Brief Title: Pharmacogenomics Results Affect Patients' Plan of Care and Changes in Medication Prescription(s)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Collaborators: PAS Research Services (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1463
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Pharmacogenomic
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: pharmacogenomic — Standard Operating Procedures on Pharmacogenomic testing and changes made to specific SOP

SUMMARY:
Current providers' standard operating procedures on pharmacogenomic testing patients

DETAILED DESCRIPTION:
The general design of this study is collecting data and reviewing Principal Investigators' Standard Operating Procedures on Pharmacogenomic testing and changes made to their specific SOP.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Medical Practitioner

  * Medical Doctor (MD)
  * Doctor of Osteopathic (DO)
  * Physician Assistant (PA)
  * Advanced Practice Registered Nurse (APRN)
  * Nurse Practioner (NP)
* Must have a current standard operating procedure that includes obtaining/reviewing medical history.

Exclusion Criteria:

* Government-funded insurance data cannot be included in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Current standard operating procedures for providers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-03-22 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Provider Structures and Processes | 36 months
  Plan of Care Changes due to Pharmacogenomic testing. Provider based observational survey system on the health and well-being of patients and populations

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided